CLINICAL TRIAL: NCT00839969
Title: A Randomized Study of Cystoscopy and Urethral Dilatation Versus Cystoscopy Alone in Women With Overactive Bladder Syndrome and Impaired Voiding.
Brief Title: Cystoscopy Plus Urethral Dilatation Versus Cystoscopy Alone in Women With Overactive Bladder Syndrome and Impaired Voiding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Mr Jonathan Duckett, Medway NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08/H1101/97
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Overactive Bladder Syndrome; Voiding Dysfunction
Keywords: overactive bladder syndrome; voiding; pressure flow studies; urethral dilatation
MeSH Terms: interventions — Cystoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cystoscopy alone (Sham Comparator): Women in this arm will undergo saline cystoscopy under general anaesthesia only.
  Interventions: Procedure: Cystoscopy
- Cystoscopy and urethral dilatation (Active Comparator): Women in this group will undergo cystoscopy and urethral dilatation under general anaesthesia
  Interventions: Procedure: Cystoscopy and urethral dilatation

INTERVENTIONS:
Procedure: Cystoscopy — Saline cystoscopy under general anaesthesia
  Arms: Cystoscopy alone
Procedure: Cystoscopy and urethral dilatation — Saline cystoscopy and urethral dilatation (using Hegar dilators) under general anaesthesia
  Arms: Cystoscopy and urethral dilatation

SUMMARY:
Urethral dilatation is a commonly undertaken intervention for a variety of urinary complaints including overactive bladder symptoms. There is however very little evidence for its efficacy, and no randomized trial evidence. The aim of this study is to ascertain the effect of urethral dilatation on overactive bladder symptoms and on voiding parameters. The null hypothesis is that there will be no difference in symptoms or voiding parameters between the urethral dilatation and sham groups.

Eligible women will be assessed initially with a history and examination, a King's Health Questionnaire and Bristol Female Urinary Tract Symptoms (BFLUTS) questionnaire and pressure flow studies. They will be randomized to undergo either cystoscopy alone or cystoscopy and urethral dilatation. Patients will be blinded to the procedure undertaken and randomized using a series of opaque envelopes. Follow up will be at 6 weeks with repeat questionnaires and pressure flow studies. Subjective and objective outcomes will be compared between the two groups.

DETAILED DESCRIPTION:
This study is a randomised controlled trial. Objective outcomes will be evaluated at 6 weeks' post-operatively. Subjective outcomes will be evaluated at 6 weeks' and 6 months' post-operatively.

Study Population Entry to the study will be offered to all women with OAB symptoms with impaired voiding on cystometry (flow rate less than 15mls/sec with volume of 200mls voided and a normal or high detrusor pressure at maximum flow), who have failed to improve with 2 different anticholinergic medications. Subjects will be recruited from the Urogynaecology clinic at Medway Maritime Hospital. A power calculation was carried out which showed a minimum sample size of 30 (i.e. 15 in each arm) to be necessary to ensure an 80% power with a significance level of 0.05.

Pre-operative Assessment All patients will undergo an initial assessment consisting of a full urogynaecogical history and examination, BFLUTS questionnaire and Urgency Perception Scale, and pressure flow studies. As mentioned before, each patient will have been treated with anticholinergic medications prior to being offered this intervention.

Surgical Technique All procedures will be carried out under general anaesthesia. A dose of intravenous gentamicin will be given to each patient at induction. After emptying the bladder, saline cystoscopy will be carried out with a 30 degree cystoscope. The bladder mucosa will be systematically inspected for any abnormalities and the bladder filled either until the sphincter mechanism is overcome or to 1000mls. The bladder is emptied again and a second fill undertaken. The bladder mucosa is inspected for petechial haemorrhages, erythema and other signs of chronic cystitis on the second fill.

In subjects randomised to undergo urethral dilatation, this will be undertaken using Hagar dilators. There is no evidence in the literature regarding normal urethral calibre in women. Therefore, the urethra will be dilated to a maximum of 10 Hagar as per our unit's protocol. Women will be discharged on the same day, if they pass urine adequately.

Post-operative Assessment Subjects will be seen in the Urogynaecology clinic at 6 weeks' post-operatively and assessed with a BFLUTS questionnaire, UPS and repeat pressure flow studies. Each patient will be assessed subjectively at 6 months' post-operatively using the symptom questionnaires.

Significance testing will be used to compare symptom scores and pressure flow parameters between each group pre- and post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. OAB symptoms (based on relevant domains of BFLUTS questionnaire and Urgency Perception Scale) which have not improved with 2 anticholinergic treatments.
2. Maximum flow rate of less than 15 ml/s on a volume voided of 200mls or more, with a normal or high detrusor pressure at maximum flow on pressure flow studies
3. Patients must be able to give informed consent for the study

Exclusion Criteria:

1. Presence of concurrent urodynamic stress incontinence
2. Patient unfit or unwilling to undergo a general anaesthetic
3. Patients with bladder pathology or haematuria of unknown origin
4. Patients with neurological disorders (as these may affect voiding)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Change in pressure flow parameters (voided volume, maximum flow rate, acceleration of flow rate and detrusor pressure at maximum flow) at 6 weeks' post-operatively. | 6 weeks
Change in symptoms as measured by the BFLUTS questionnaire and Urgency Perception Scale at 6 weeks' and 6 months' post-operatively. | 6 weeks and 6 months

SECONDARY OUTCOMES:
Change in quality of life status as determined by change in King's Health Questionnaire scoring at 6 weeks and 6 months' post-operatively. | 6 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Duckett, FRCOG, Principal Investigator — Medway NHS Trust
Locations (1):
- Medway Maritime Hospital, Gillingham, Kent, United Kingdom

REFERENCES:
- [Derived] Basu M, Khullar V, Duckett J. Urethral dilatation: Is there any benefit over cystoscopy and distension? A randomized trial in women with overactive bladder symptoms. Neurourol Urodyn. 2014 Mar;33(3):283-8. doi: 10.1002/nau.22411. Epub 2013 May 1. PMID 23636866